# **Cover Page**

# **Study title:**

Insertion of a Transoesophageal Echocardiography Probe Using the McGRATH Video Laryngoscope in Cardiac Surgery Patients: A Randomized Controlled Trial

### **Document Type:**

Study Protocol and Statistical Analysis Plan

### **ClinicalTrials.gov Identifier:**

NCT number not yet assigned

#### **Protocol Version Date:**

January 7, 2026

### **Investigators:**

Hassan Mohamed Ali, Cairo University

Ahmed Abdalwahab, Prince Sultan Cardiac Center

Ahmed Abuzaid, Prince Sultan Cardiac Center

## **Location and Expected Duration of the Study:**

Location: Prince Sultan Cardiac Center, Riyadh, Saudi Arabia

Cairo University, Cairo, Egypt

Expected Duration: From January 2026 to June 2026

### RESEARCH PROPOSAL

# **Project Summary**

Transoesophageal echocardiography (TEE) is an essential intraoperative monitoring tool in cardiac anesthesia. Despite its utility, TEE probe insertion can cause complications such as oropharyngeal injuries and esophageal perforation. Reported rates of oropharyngeal injury range from 0.2% to 1.2%, and esophageal perforation occurs in 0.01% to 0.09% of patients. Most injuries are located at the upper esophagus, particularly near the esophageal inlet. Assisting probe insertion using a conventional Macintosh laryngoscope has been suggested to reduce such injuries. However, its limited visualization of the esophageal inlet remains a challenge. The McGRATH video laryngoscope provides a superior view of upper airway anatomy, including the glottis and esophageal inlet, and may therefore offer safer and more efficient TEE probe placement.

# **Project Objectives**

Primary objectives:

•To compare the incidence of pharyngeal mucosal injury during TEE probe insertion between patients using the McGRATH video laryngoscope and those using the Macintosh laryngoscope.

Secondary Objectives:

• To compare the visibility of the oesophageal inlet during insertion.

- To measure the duration of TEE probe insertion.
- To assess the number of insertion attempts.

### Literature Survey/Background

Although transoesophageal echocardiography (TEE) is considered a well tolerated technique, rare but serious complications have been reported.[1-6] In anaesthetised patients, the total incidence of oropharyngeal injury associated with insertion of a TEE probe ranges from 0.2 to 1.2%,[1,3,5] and orogastric tract perforation, the most feared complication, occurs in 0.01 to 0.09% of both ambulatory and anaesthetized patients.[1-4] When orogastric tract perforation occurs, it most commonly affects the hypopharynx and the oesophagus, the incidence of which are 0.01 and 0.02%, respectively.[7-9] Oesophageal perforation occurs more frequently in the upper oesophagus including the oesophageal inlet than in the middle to lower oesophagus. [1,2,4] This is probably because the crossing of fibres from the constrictor muscle of the pharynx and the cricopharyngeus muscle make this portion of the oesophagus particularly susceptible to injury and perforation.[4] The incidence of minor adverse effects related to TEE probe insertion such as oropharyngeal mucosal injury seems to be more frequent in anaesthetized patients, but data is lacking and there is just a single study that puts the incidence of mucosal injury after blind TOE probe insertion at 55%, a relatively high figure.[10] Perforation of the hypopharynx and upper oesophagus after TEE probe insertion is likely to be caused by difficulties introducing the probe into the inlet of the oesophagus, generating undue pressure at the tip of the probe. Mucosal injury in the pharynx and oesophageal inlet per se is not serious but would also result from excessive pressure exerted by the probe tip. Prevention of these complications requires that force during insertion is avoided, and for this, direct visualization of the inlet of the oesophagus is desirable. Insertion under direct vision with a Macintosh laryngoscope (Macintosh) can reduce the high incidence of oropharyngeal injury from 55 to 5%.[10] The presence of an endotracheal tube prevents direct visualisation of the oesophageal inlet even when using the Macintosh, and it may sometimes be difficult to observe the passage of a TEE probe, creating conditions for pharyngeal injury.

The McGRATH MAC (McGRATH; Aircraft Medical Ltd., Edinburgh, UK) is a video laryngoscope that provides a better view of the glottis, piriform fossa and oesophageal inlet in tracheal intubation than the Macintosh.[11,12] We hypothesize

that the McGRATH will provide better visualization of the oesophageal inlet and will reduce the incidence of pharyngeal injury related to insertion of a TEE probe.

### **Research Design**

Prospective, randomized controlled study

#### Methods

This study will be conducted between January 2026 and June 2026. Written informed consent will be obtained from each patient, who will agree to be enrolled in the study.

Inclusion criteria:

- Adults (male or female), aged above 18
- ASA physical status II or III
- Scheduled for elective cardiac surgery under general anesthesia requiring intraoperative TEE
- Provide written informed consent

Exclusion criteria:

Patients with any of the following will be excluded:

- •Dysphagia or sore throat
- •oropharyngeal infection
- •cervical spine pathology

# Randomization and group allocations:

Randomization will be done by online random number generator software (https://www.sealedenvelope.com/simple-randomiser/v1/lists) into either a Macintosh (C group) or a McGRATH (M group) group using blocks of random sizes of 4. The group allocations will be contained in sealed envelopes that will be opened in the operating theatre suite after the enrolment procedure had been completed.

Three cardiac anaesthesiologists with more than 5 years of experience intraoperative TEE will participate in this study and will insert the TEE probe.

All patients will be assessed preoperatively using the Mallampati classification, and after induction of general anesthesia; the patients of both groups will have tracheal intubation. TEE probe assisted insertion with Macintosh or McGRATH will be done with the patient head in neutral position. External laryngeal manipulation and repositioning of the blade will not be allowed in the first trial. The esophageal inlet visibility will be assessed, and the time of insertion will be recorded.

#### **Measurements:**

The endpoints will include: each patient's demographics, Mallampati classification (MP), esophageal inlet visibility, numbers of insertion trials, duration for TEE probe insertion, vital signs pre and during the insertion (heart rate, blood pressure, and oxygen saturation), and presence of complications after removal of the probe and anesthesiologist satisfaction.

We defined the duration of TEE probe insertion as the time, measured in seconds, from the moment the mouth will be opened until the TEE probe will be fully inserted. The range of a single trial will be delineated from the insertion of the TEE probe into the mouth to its removal or insertion into the esophagus. The total time for TEE probe manipulation will be calculated by summing the durations of multiple trials, excluding the intervals between manipulations. We will evaluate pharyngeal injury as a trauma-related factor. Pharyngeal injury will be defined as observation of laceration and/or hematoma with the McGRATH after the TEE probe has been removed by a blinded observer to the group allocation. Also, he will record the presence or absence of laceration and/or hematoma in the posterior pharyngeal wall, postcricoid area, lateral and medial wall of the piriform sinus and the inlet area to the esophagus.

## **Sample size Calculation:**

A preliminary study (internal data) showed:

- Visibility of oesophageal inlet: 40% (Macintosh) vs. 80% (McGRATH)
- Pharyngeal injury: 2% (Macintosh) vs. 0.7% (McGRATH)

To detect a reduction in mucosal injury from 2% to 0.7% with 80% power and alpha = 0.05, 50 patients per group (total n = 100) are required.

#### Statistical analysis

The Shapiro–Wilk test will be used to assess continuous variables for normality. Normally distributed continuous data will be analyzed by Student's t test. The Mann-Whitney U test will be used for analysis of the number of TEE insertion attempts. The x2 test will be used for analysis of the incidence of pharyngeal mucosal injury and visibility of the oesophageal inlet. All analyses will be performed using GraphPad Prism version 6.0 (GraphPad Software, San Diego, California, USA). Data will be presented as mean ±SD. A P value less than 0.05 will be considered statistically significant.

### **Interim Analysis and Safety Monitoring**

An interim safety analysis will be conducted after 50 patients (50% enrolment). The study will be paused if:

- The rate of mucosal injury in either group exceeds 25%
- A statistically significant increase in complications is detected by The Data Safety Monitoring Board (DSMB) will review interim results and recommend continuation, modification, or early termination. The study will follow an intention-to-treat analysis approach.

#### **Ethical Considerations**

- Informed consent will be obtained from all participants.
- Confidentiality will be maintained in accordance with institutional and national standards.
- Adverse events will be recorded and reported promptly to the IRB.
- No financial compensation or inducements will be provided to participants.

#### References

- [1] Kallmeyer IJ, Collard CD, Fox JA, et al. The safety of intraoperative transesophageal echocardiography: a case series of 7200 cardiac surgical patients. Anesth Analg 2001; 92:1126–1130.
- [2] Min JK, Spencer KT, Furlong KT, et al. Clinical features of complications from transesophageal echocardiography: a single-center case series of 10,000 consecutive examinations. J Am Soc Echocardiogr 2005; 18:925–929.
- [3] Lenon MJ, Gibbs NM, Weightman WM, et al. Transesophageal echocardiography-related gastrointestinal complications in cardiac surgical patients. J Cardiothorac Vasc Anesth 2005; 19:141–145.
- [4] Bavalia N1, Anis A, Benz M, et al. Esophageal perforation, the most feared complication of TEE: early recognition by multimodality imaging. Echocardiography 2011; 28:E56–E59.
- [5] Piercy M,McNicol L, Dinh DT, et al. Major complications related to the use of transesophageal echocardiography in cardiac surgery. J Cardiothorac Vasc Anesth 2009; 23:62–65.
- [6] Kharasch E, Sivarajan M. Gastroesophageal perforation after intraoperative transesophageal echocardiography. Anesthesiology 1996; 85:426–428.
- [7] Spahn DR, Schmid S, Carrel T, et al. Hypopharynx perforation by a transesophageal echocardiography probe. Anesthesiology 1995; 82:581–583.
- [8] BakhosD,Cottier JP, Beutter P, Morinie're S. Hypopharyngeal perforation: an unusual complication of transesophageal echocardiography. Ear Nose Throat J 2011; 90:E1–E2.
- [9] Aviv JE, Di Tullio MR, Homma S, et al. Hypopharyngeal perforation near-miss during transesophageal echocardiography. Laryngoscope 2004; 114:821–826.
- [10] Na S, Kim CS, Kim JY, et al. Rigid laryngoscope-assisted insertion of transesophageal echocardiography probe reduces oropharyngeal mucosal injury in anesthetized patients. Anesthesiology 2009; 110:38–40.
- [11] Noppens RR, Mobus S, Heid F, et al. Evaluation of the McGrath Series 5 videolaryngoscope after failed direct laryngoscopy. Anaesthesia 2010; 65:716–720.

[12] Shippey B, Ray D, McKeown D. Use of the McGrath1 videolaryngoscope in the management of difficult and failed tracheal intubation. Br J Anaesth 2008; 100:116–119.